CLINICAL TRIAL: NCT01832662
Title: Coffee Antioxidant Efficacy in Humans
Brief Title: Coffee Polyphenols Antioxidants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 10.07.MET
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
MeSH Terms: interventions — Coffee; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Coffee (Experimental): 4 cups/day of 2.5g of coffee each
  Interventions: Other: coffee polyphenols mixed with placebo; Other: maltodextrin enriched with caffeine
- coffee polyphenols mixed with placebo (Active Comparator): 4 cups/day of 2.5g of product each
  Interventions: Other: coffee; Other: maltodextrin enriched with caffeine
- maltodextrin enriched with caffeine (Placebo Comparator): 4 cups/day of 2.5g of product each
  Interventions: Other: coffee; Other: coffee polyphenols mixed with placebo

INTERVENTIONS:
Other: coffee — coffee, placebo enriched with polyphenols and placebo with caffeine
  Arms: coffee polyphenols mixed with placebo; maltodextrin enriched with caffeine
Other: coffee polyphenols mixed with placebo — coffee polyphenols mixed with placebo
  Arms: Coffee; maltodextrin enriched with caffeine
Other: maltodextrin enriched with caffeine — maltodextrin enriched with caffeine
  Arms: Coffee; coffee polyphenols mixed with placebo

SUMMARY:
Coffee is one of the most widely consumed beverages. It contains polyphenols (chlorogenic acids) and bioavailability of these bioactive compounds is now somewhat well understood. In addition, chlorogenic acids are known to be antioxidants in the cup, but reliable evidence remains to be observed in vivo. The objective of this trial is to understand if regular (10d) coffee intake may be beneficial on biomarkers of oxidative damage measured in urine and plasma. A secondary objective is to understand if polyphenols isolated from coffee may be as beneficial as the whole beverage in reducing oxidative stress compared to placebo

DETAILED DESCRIPTION:
This is an interventional study with a crossover randomized placebo-controlled double-blind design to assess the effect of regular consumption of coffee on oxidative stress compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 70 years, male and female
* healthy
* BMI 19 - 29 kg/m2
* Coffee drinkers with an average consumption of 1-3 cups per day
* having given informed consent

Exclusion Criteria:

* Intestinal or metabolic diseases / disorders such as diabetic, renal, hepatic, hypertension, pancreatic or ulcer- Have had a gastrointestinal surgery, except appendicectomy
* Difficulty to swallow
* Have a regular consumption of medication
* Have taken antibiotic therapy within the last 6 months
* Alcohol consumption > 2 units a day
* Smokers (more than 5 cigarettes per day)
* Have given blood within the last 3 weeks
* Volunteers who cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial during the last 3 weeks

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
oxidative stress | Change in plasma and in urine beta isoprostane from baseline to the last day of a 10-day period of product intake
  The level of oxidative stress will be assessed through measurements of urine and plasma beta isoprostane

SECONDARY OUTCOMES:
bioavailability of coffee phenolics | Change of plasma chrorogenic and phenolic acids from baseline to the last day of a 10-day period of product intake
  plasma kinetics of chlorogenic and phenolic acids.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, Principal Investigator — Nestlé Clinical Development Unit